CLINICAL TRIAL: NCT03552562
Title: Measurement of Total Retinal Blood Flow and Oxygen Extraction in Patients With Diabetes and Healthy Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv.-Doz. Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: OPHT-100218
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Retinal Blood Flow

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 30 patients with no signs of diabetic retinopathy (Other)
  Interventions: Device: Fourier Domain Color Doppler Optical Coherence Tomography (FDOCT)
- 30 patients with mild diabetic retinopathy (Other)
  Interventions: Device: Fourier Domain Color Doppler Optical Coherence Tomography (FDOCT)
- 30 patients with moderate to severe diabetic retinopathy (Other)
  Interventions: Device: Fourier Domain Color Doppler Optical Coherence Tomography (FDOCT)
- 30 healthy age-and sex- matched control subjects (Other)
  Interventions: Device: Fourier Domain Color Doppler Optical Coherence Tomography (FDOCT)

INTERVENTIONS:
Device: Fourier Domain Color Doppler Optical Coherence Tomography (FDOCT) — Fourier domain OCT is based on a local phase analysis of the backscattered signal and allows for bidirectional Doppler flow imaging.(Leitgeb et al. 2003a; Leitgeb et al. 2003b) It does not need reference arm scanning and records one full depth and Doppler profile in parallel. The system operates with an equivalent A-scan rate of 25 kHz and allows real time imaging of the color encoded Doppler information together with the tissue morphology at a rate of 2-4 tomograms (40 x 512 pixel) per second. Despite the high detection speed we achieve a system sensitivity of 86dB using a beam power of 500μW at the cornea. The fundus camera allows simultaneous view for selection of the region of interest. We observe bi-directional blood flow and pulsatility of blood velocity in retinal vessels with a Doppler detection bandwidth of 12.5 kHz and a longitudinal velocity sensitivity in tissue of 200μm/s. Diffuse luminance flicker will be applied during the measurements for 60 seconds.

SUMMARY:
The prevalence of diabetes and diabetes-associated complications is still increasing. Several major long-term complications of diabetes such as cardiovascular disease, chronic renal failure, diabetic retinopathy and others relate to the damage of blood vessels. Given that the eye provides the unique possibility in the human body to directly visualize blood vessels, much interest has been directed towards studying the ocular circulation and retinal oxygen metabolism.

Although data of large epidemiological studies indicate that changes in retinal vessel caliber reflect other diabetes related factors, such as fasting glucose levels, there is still conflicting evidence on blood flow alterations in patients with diabetes. Strongly related to ocular blood flow, investigation of retinal oxygen metabolism has received a lot attention. In particular, hypoxia is assumed to be major trigger of neovascularisation in the retinal of diabetic patients The present study seeks to investigate both ocular blood flow and tissue oxygen extraction in patients with type II diabetes. For this purpose, total retinal blood flow will be assessed with bi-directional Fourier Domain Doppler Optical Coherence Tomography (FDOCT). Furthermore, retinal oxygen saturation will be measured non-invasively by a fundus camera based system. Based on data of retinal blood flow and retinal oxygen saturation, retinal oxygen. This will help to better understand ocular blood flow changes and oxygen metabolism in patients with type II diabetes.

ELIGIBILITY:
Inclusion Criteria for healthy subjects:

* Men and women aged over 18 years
* Non-smokers
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 6 Dpt.

Inclusion criteria for patients with diabetes

* Men and women aged over 18 years
* Non-smokers
* Previously diagnosed type II diabetes
* No, mild, moderate or severe non-proliferative diabetic retinopathy
* Normal ophthalmic findings except mild diabetic retinopathy, ametropy < 6 Dpt.

Exclusion Criteria for healthy subjects:

* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition as judged by the clinical investigator
* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study (except oral contraceptive)
* untreated arterial hypertension (defined as either systolic blood pressure >145 mmHg or diastolic blood pressure >90 mmHg)
* Blood donation during the previous three weeks
* History or family history of epilepsy
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Best corrected visual acuity < 0.8 Snellen
* Ametropy ≥ 6 Dpt
* Pregnancy, planned pregnancy or lactating

Exclusion Criteria for patients with diabetes:

* Participation in a clinical trial in the 3 weeks preceding the screening visit
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition, except diabetes, as judged by the clinical investigator
* untreated arterial hypertension (defined as either systolic blood pressure >145 mmHg or diastolic blood pressure >90 mmHg)
* Blood donation during the previous three weeks
* Moderate to severe non-proliferative or proliferative diabetic retinopathy
* Previous laser photocoagulation treatment
* History or family history of epilepsy
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Best corrected visual acuity < 0.8 Snellen
* Ametropy ≥ 6 Dpt
* Pregnancy, planned pregnancy or lactating

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
Total retinal blood flow (DVA and FDOCT) | 60 minutes
  To determine the total blood flow in the eye, OCT measurements were performed with a rectangular scanning pattern around the optical nerve head.

OTHER OUTCOMES:
Retinal vessel diameter (DVA) | 30 minutes
  The DVA allows for the real time measurement of retinal vessel diameters in vivo.
  The DVA is a commercially available system (IMEDOS, Jena, Germany) which comprises a fundus camera, a video camera, a real time monitor and a personal computer with an analyzing software for the accurate determination of retinal arterial and venous diameters. Every second a maximum of 25 readings of vessel diameter can be obtained. For this purpose the fundus is imaged onto the charge coupled device chip of the video camera. The consecutive fundus images are digitized using a frame grabber. In addition, the fundus image can be inspected on the real time monitor and, if necessary, stored on a video recorder. Evaluation of the retinal vessel diameters can either be done online or offline from the recorded video tapes
Retinal oxygen saturation (DVA) | 30 minutes
  In particular, retinal oxygen saturation measurement is based on the image analysis by the DVA software of two monochromatic fundus images as recorded by a standard DVA. In an image, obtained by the camera and filter assembly, the operator has to mark the vessel of interest by a mouse click. The vessel is traced automatically applying the following procedure. The vessel walls are located as photometric edges in the vicinity of the mouse cursor in the green channel image. If edges are determined, the search is continued in their proximity.
Retinal blood velocities (FDOCT) | 15 minutes
  We observe bi-directional blood flow and pulsatility of blood velocity in retinal vessels with a Doppler detection bandwidth of 12.5 kHz and a longitudinal velocity sensitivity in tissue of 200μm/s.
Blood flow response of retinal vessels to increased neuronal activity Ocular perfusion pressure | 30 minutes
Retinal nerve fiber layer thickness (OCT) | 15 minutes
  Peripapillary retinal nerve fiber thickness will be assessed using a commercially available device (Heidelberg Spectralis).
Central retinal thickness (OCT) | 5 minutes
  Central retinal thickness will be assessed using a commercially available device (Heidelberg Spectralis).
Pattern Electroretinography (pERG) | 15 minutes
  Pattern ERG will be performed according to the ISCEV standard for clinical pattern Electroretinography. Briefly described, the gold wire will be placed in a lower conjunctival sac, attached to the lateral nasal surface on one site and covered by the gold foil electrode on the temporal site. Reference and the ground electrodes will be placed in the outer canthus and the forehead, respectively. A black-and-white reverse checkerboard will be used with an aspect ratio of the width over the height of the stimulus field not exceeding 4:3.
Capillary blood glucose level | 5 minutes
  Capillary blood glucose levels will be measured using a commercially available glucose meter (Accu- Check Go, Roche Diagnostics GmbH, Vienna). Capillary blood will be sampled from one fingertip with a single-use lancet.
Oxygen and carbon dioxide partial pressure in arterialized blood | 10 minutes
  The arterialized blood will be drawn into a thin glass capillary tube. Arterial pH, pCO2 and pO2 will be determined with an automatic blood gas analysis system (AVL 995-Hb, Graz, Austria).
Autonomic and sensomotoric neuropathy measurements | 30 minutes
  Assesment of heart rate variability is a standardized, non invasive method for quantification of autonomic (sympathetic and parasympathetic) control and thus preferably used for evaluation of cardiovascular autonomic neuropathy (CAN) in diabetes. This measurement of CAN is based on analysis of heart rate variability either in time-domain (cardiovascular reflex tests to standardized stimuli including deep breathing, Valsalva maneuver and orthostatic load)or in frequency-domain, using a short-term modified orthostatic load. Short- term spectral analysis of HRV is obtained from recordings consisting of 256 seconds of artifact-free records each using a VariaCardio® system (Advanced Medical Diagnostics Group, UK).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Austria, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No